CLINICAL TRIAL: NCT04651088
Title: Evaluation of Multiple Alkalinizing Agents on Urinary Stone Risk Parameters in Stone and Non-stone Formers on a Metabolically Controlled Diet
Brief Title: Comparing Alkalinizing Agents Efficacy on Stone Risk in Patients on a Metabolically Controlled Diet
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Brett Johnson, Associate Professor of Urology, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STU-2020-0613
Record Dates: First submitted 2020-11-04; First posted 2020-12-03 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Kidney Stone
MeSH Terms: conditions — Kidney Calculi | interventions — Potassium Citrate; Sodium Bicarbonate; potassium bicarbonate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Metabolic diet (Placebo Comparator): Controlled metabolic diet arm.
  Interventions: Drug: Potassium citrate; Drug: Sodium bicarbonate; Dietary Supplement: Litholyte; Dietary Supplement: Crystal Lite; Drug: Potassium Bicarbonate
- Potassium citrate (Active Comparator)
  Interventions: Drug: Potassium citrate; Drug: Sodium bicarbonate; Dietary Supplement: Litholyte; Dietary Supplement: Crystal Lite; Drug: Potassium Bicarbonate
- Sodium Bicarbonate (Active Comparator)
  Interventions: Drug: Potassium citrate; Drug: Sodium bicarbonate; Dietary Supplement: Litholyte; Dietary Supplement: Crystal Lite; Drug: Potassium Bicarbonate
- Litholyte arm (Active Comparator)
  Interventions: Drug: Potassium citrate; Drug: Sodium bicarbonate; Dietary Supplement: Litholyte; Dietary Supplement: Crystal Lite; Drug: Potassium Bicarbonate
- Crystal Lite (Active Comparator)
  Interventions: Drug: Potassium citrate; Drug: Sodium bicarbonate; Dietary Supplement: Litholyte; Dietary Supplement: Crystal Lite; Drug: Potassium Bicarbonate
- Potassium Bicarbonate (Active Comparator)
  Interventions: Drug: Potassium citrate; Drug: Sodium bicarbonate; Dietary Supplement: Litholyte; Dietary Supplement: Crystal Lite; Drug: Potassium Bicarbonate

INTERVENTIONS:
Drug: Potassium citrate — Slow release potassium citrate UroCit-K. Participants will take 20mEq twice daily.
Drug: Sodium bicarbonate — 650mg tabs. Take 3 tabs twice daily.
Dietary Supplement: Litholyte — One packet is taken with 170ml of water. Two packets daily.
Dietary Supplement: Crystal Lite — The classic lemonade contains 21.7mEq/liter of alkali Therefore, patients will take 2 litres daily to have the 40mEq of alkali daily needed.
Drug: Potassium Bicarbonate — 20 mEq tablets, one tablet twice daily

SUMMARY:
The purpose of this study is to compare over the counter and alternative prescription urinary alkalinizing agents to slow release potassium citrate in their ability to modify urinary parameters associated with stone formation.

DETAILED DESCRIPTION:
Kidney stones are a common medical problem, occurring in almost 10% of people in the United States1. Furthermore, 50% of patients will recur within 10 years2. Metabolic testing is advised in recurrent stone formers, as well as those considered high risk, to assess for a specific abnormality which may prompt intervention to prevent future stone formation. Non-surgical interventions include both dietary counselling, as well as pharmacotherapy.

One of the most commonly prescribed class of pharmacotherapies is alkali therapy which can be used to both increase the urinary pH and raise the urine citrate levels. This is particularly useful as correction of very acidic urinary pH (<5.5) can counteract uric acid crystallization thereby preventing or even dissolving uric acid stones3. Further, citrate has been shown to be a potent inhibitor of calcium stones by binding to the calcium directly4 and inhibiting crystal nucleation, thereby reducing calcium stone formation5,6.

The most commonly utilized preparation of alkali therapy is potassium citrate which has been shown to prevent stone formation better than sodium citrate7. Unfortunately, some forms of potassium citrate (crystal packets) have become unavailable, and the slow release form of potassium citrate (UroCit-K) now exceeds $15/day in cost8. There have been multiple alternative alkali therapies that have been used in place of potassium citrate, including both medical foods and prescription medications, but with little evidence to support their use. A pilot study in order to quantify the metabolic effects of these agents and compare them to potassium citrate will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and older.
* with or without a history of stone disease.

Exclusion Criteria:

* They are unable to take any of the medications due to health reasons.
* Participants are pregnant or nursing.
* Participants are unable to adhere to the metabolic diet.
* Participants had a prior adverse event from one or more of the medications.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
24 hour urine volume | Change from baseline (Day 4) to initial start on treatment (Day 5)
  Total urine volume
24 hour urine volume | Change from baseline (Day 4) to end of study (day 12)
  Total urine volume
24 hour urine creatinine | Change from baseline (Day 4) to initial start on treatment (Day 5)
  Urine creatinine
24 hour urine creatinine | Change from baseline (Day 4) to end of study (day 12)
  Urine creatinine
24 hour urine calcium | Change from baseline (Day 4) to initial start on treatment (Day 5)
  urine calcium
24 hour urine calcium | Change from baseline (Day 4) to end of study (day 12)
  urine calcium
24 hour urine potassium | Change from baseline (Day 4) to initial start on treatment (Day 5)
  Urine potassium
24 hour urine potassium | Change from baseline (Day 4) to end of study (day 12)
  Urine potassium
24 hour urine sodium | Change from baseline (Day 4) to initial start on treatment (Day 5)
  Urine sodium
24 hours urine sodium | Change from baseline (Day 4) to end of study (day 12)
  Urine sodium
24 hours urine citrate | Change from baseline (Day 4) to initial start on treatment (Day 5)
  Urine citrate
24 hours urine citrate | Change from baseline (Day 4) to end of study (day 12)
  Urine citrate
24 hours urine uric acid | Change from baseline (Day 4) to initial start on treatment (Day 5)
  Urine uric acid
24 hours urine uric acid | Change from baseline (Day 4) to end of study (day 12)
  Urine Uric Acid
24 hours urine oxalate | Change from baseline (Day 4) to initial start on treatment (Day 5)
  Urine oxalate
24 hours urine oxalate | Change from baseline (Day 4) to end of study (day 12)
  Urine oxalate
24 hours urine magnesium | Change from baseline (Day 4) to initial start on treatment (Day 5)
  Urine magnesium
24 hours urine magnesium | Change from baseline (Day 4) to end of study (day 12)
  Urine magnesium
24 hours urine ammonia | Change from baseline (Day 4) to initial start on treatment (Day 5)
  Urine ammonia
24 hours urine ammonia | Change from baseline (Day 4) to end of study (day 12)
  Urine ammonia
24 Hour Urine pH | Change from baseline (Day 4) to initial start on treatment (Day 5)
  Overal Urine pH from 24h urine sample.
24 Hour Urine pH | Change from baseline (Day 4) to end of study (day 12)
  Overal Urine pH from 24h urine sample.
24 hour urine phosphorus | Change from baseline (Day 4) to initial start on treatment (Day 5)
  Urine phosphorus
24 hour urine phosphorus | Change from baseline (Day 4) to end of study (day 12)
  Urine phosphorus
24 hour urine sulfate | Change from baseline (Day 4) to initial start on treatment (Day 5)
  Urine sulfate
24 hour urine sulfate | Change from baseline (Day 4) to end of study (day 12)
  Urine sulfate

SECONDARY OUTCOMES:
# of patient who adherence to 100% Medication | At the end of study approximately 10 weeks after start of study.
  Patient's adherence to medication for duration of study.
Total out of pocket cost | At the end of study approximately 10 weeks after start of study.
  Calculate and compare treatment costs for the different interventions (in American dollars).
Patient's Satisfaction Survey | At the end of study approximately 10 weeks after start of study.
  Patient satisfaction survey, adapted from the Treatment Satisfaction Questionnaire for Medication-14. Patients are queried on their satisfaction, with 9 questions for each medication.
Patient's GI Distress | At the end of study approximately 10 weeks after start of study.
  Patient's GI distress symptom scale measures patients GI distress. There are 18 questions with descriptive answers ranging from "none", "mild", "moderate", "quite a lot" and "unbearable". There are no numerical scores, rather just descriptive scores. "None" means no GI distress, "unbearable" means that you are in a lot of distress from your GI symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scales CD Jr, Smith AC, Hanley JM, Saigal CS; Urologic Diseases in America Project. Prevalence of kidney stones in the United States. Eur Urol. 2012 Jul;62(1):160-5. doi: 10.1016/j.eururo.2012.03.052. Epub 2012 Mar 31. PMID 22498635
- [Background] Uribarri J, Oh MS, Carroll HJ. The first kidney stone. Ann Intern Med. 1989 Dec 15;111(12):1006-9. doi: 10.7326/0003-4819-111-12-1006. PMID 2688503
- [Background] Pearle MS, Goldfarb DS, Assimos DG, Curhan G, Denu-Ciocca CJ, Matlaga BR, Monga M, Penniston KL, Preminger GM, Turk TM, White JR; American Urological Assocation. Medical management of kidney stones: AUA guideline. J Urol. 2014 Aug;192(2):316-24. doi: 10.1016/j.juro.2014.05.006. Epub 2014 May 20. PMID 24857648
- [Background] Pak CY, Sakhaee K, Fuller C. Successful management of uric acid nephrolithiasis with potassium citrate. Kidney Int. 1986 Sep;30(3):422-8. doi: 10.1038/ki.1986.201. PMID 3784284
- [Background] Ryall RL. Urinary inhibitors of calcium oxalate crystallization and their potential role in stone formation. World J Urol. 1997;15(3):155-64. doi: 10.1007/BF02201852. No abstract available. PMID 9228722
- [Background] Preminger GM, Sakhaee K, Skurla C, Pak CY. Prevention of recurrent calcium stone formation with potassium citrate therapy in patients with distal renal tubular acidosis. J Urol. 1985 Jul;134(1):20-3. doi: 10.1016/s0022-5347(17)46963-1. PMID 4009822
- [Background] Ettinger B, Pak CY, Citron JT, Thomas C, Adams-Huet B, Vangessel A. Potassium-magnesium citrate is an effective prophylaxis against recurrent calcium oxalate nephrolithiasis. J Urol. 1997 Dec;158(6):2069-73. doi: 10.1016/s0022-5347(01)68155-2. PMID 9366314
- [Background] Preminger GM, Sakhaee K, Pak CY. Alkali action on the urinary crystallization of calcium salts: contrasting responses to sodium citrate and potassium citrate. J Urol. 1988 Feb;139(2):240-2. doi: 10.1016/s0022-5347(17)42374-3. PMID 3339718
- [Background] Stern KL, Canvasser N, Borofsky M, Gleason VM, Kamphuis G, El Tayeb MM, Hsi R, Scotland KB. Alkalinizing Agents: A Review of Prescription, Over-the-Counter, and Medical Food Supplements. J Endourol. 2020 Jan;34(1):1-6. doi: 10.1089/end.2019.0292. Epub 2019 Sep 25. PMID 31333065